CLINICAL TRIAL: NCT00108498
Title: New Pharmacological Treatment for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RESP-011-02F
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; mirtazapine; sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Mirtazapine

INTERVENTIONS:
Drug: mirtazapine

SUMMARY:
This study will determine if mirtazapine, a unique antidepressant that does not disturb sleep, will improve obstructive sleep apnea (OSA). The design is randomized, crossover, double blind, and placebo controlled. On two consecutive nights of one week, the patients receive either 30 mg mirtazapine or placebo at bedtime. The following week, the alternative medication is administered. The patients have known mild to moderate sleep apnea. The endpoints of the study are the apnea + hypopnea index (AHI), sleep quality, and the degree of arterial oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Known OSA mild to moderate

Exclusion Criteria:

* On antidepressant or antipsychotic medications

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2007-03

PRIMARY OUTCOMES:
The apnea + hypopnea index (AHI)
Sleep quality
The degree of arterial oxygen desaturation

CONTACTS AND LOCATIONS:
Locations (1):
- Malcom Randall VAMC, Gainesville, Florida, United States